CLINICAL TRIAL: NCT02816138
Title: Depressed Mood Improvement Through Nicotine Dosing (Depressed MIND Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Warren Taylor, Associate Professor of Psychiatry, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DepMIND
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Major Depressive Disorder
Keywords: Geriatrics; Depression; Elderly; Cognition; Memory
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal nicotine patch (Experimental): Transdermal nicotine patch, administered on awakening and removed at bedtime (16h/d). Dosing 3.5mg patch/daily, titrated over study to maximum dose of 21mg patch/daily.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Open-label transdermal nicotine patch
  Other Names: Nicotrol; Nicoderm CQ

SUMMARY:
Late-life depression is characterized by both affective (mood) symptoms and cognitive deficits. There is currently no intervention that may provide consistent benefits to both mood and cognitive performance. Agonist activity at the nicotinic acetylcholine receptors via transdermal nicotine patches may provide benefit to both mood and cognition, working through nicotine's effects on brain neural networks, specifically the cognitive control network and default mode network.

In this initial pilot project, the investigators will test this hypotheses in 15 nonsmoking depressed elders with subjective cognitive impairment. Following baseline neuroimaging and cognitive testing, participants will receive 12 weeks of open-label transdermal nicotine. Afterwards, participants will repeat neuroimaging and cognitive assessments.

DETAILED DESCRIPTION:
Late-life depression (LLD) is characterized both by affective symptoms and cognitive deficits. The co-occurrence of cognitive deficits in LLD is a clinically relevant phenotype characterized by significant disability and poor antidepressant response. Cognitive deficits can persist even with successful antidepressant treatment and increase the risk of depression relapse. Despite the clinical importance of cognitive deficits in LLD, there are no established treatments that specifically target cognition in this population. The lack of treatments that improve cognitive deficits in depression is a deficiency in current therapeutics.

Modulation of the cholinergic system by nicotinic receptor stimulation may improve both mood and cognition in depressed elders. Clinically, transdermal nicotine improves mood in smokers and a placebo-controlled pilot trial in nonsmoking adults found that transdermal nicotine significantly improved mood. In a previous trial examining Mild Cognitive Impairment, transdermal nicotine safely improved cognitive function on tests of attention, episodic memory, and processing speed. These same cognitive domains are impaired in LLD. The investigators hypothesize that these effects on mood and cognition are mediated through nicotine's effect to increase cognitive control network activity and reduce default mode network (DMN) activity. This pattern of network activity during tasks demanding external attention is associated with better task performance. Furthermore, as seen in smokers, nicotine's effect on these networks reduces depression's bias to negatively valenced stimuli and decreases rumination.

The central hypothesis is that in LLD, transdermal nicotine will safely improve depression by increasing activity in cognitive control regions and decreasing activity in DMN regions. This will result in a decreased attentional bias to and reactivity to negative stimuli. A secondary hypothesis is that transdermal nicotine will also improve subjective and objective cognitive performance through these same network effects.

Primary Aim 1: To determine whether administration of transdermal nicotine over 12 weeks improves clinical symptoms in patients with LLD with subjective cognitive impairment (SCI).

Hypothesis 1: Transdermal nicotine administration will result in reductions in depression severity measured by the Montgomery-Asberg Depression Rating Scale (MADRS; primary mood outcome). It will also result in improvement in broader assessments of depressive symptomatology, including anhedonia, apathy, fatigue, sleep, and rumination (secondary outcomes).

Hypothesis 2: Transdermal nicotine administration will result in improvements in attentional performance on the Conner's Continuous Performance Task (CPT; primary cognitive outcome). It will also result in improvement in subjective and objective cognitive performance on other tasks measuring attention, episodic memory, working memory, processing speed, and executive function (secondary outcomes).

Secondary Aim 2: To determine whether administration of transdermal nicotine over 12 weeks modulates canonical intrinsic functional network activity in LLD with SCI.

Hypothesis 3: On repeat administration of the Posner task of external attention, transdermal nicotine administration will result in increased activity within the cognitive control network and decreased activity within the default mode network.

Hypothesis 4: Transdermal nicotine administration will result in increased functional connectivity within the cognitive control network and decreased connectivity within the default mode network at rest.

Hypothesis 5: Changes in intrinsic network activity / connectivity with transdermal nicotine administration will be associated with changes in mood symptoms and subjective and objective cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years;
* DSM-5 (Diagnostic and statistical manual-5) diagnosis of major depressive disorder, single or recurrent episode;
* Subjective cognitive decline, defined as endorsing 20% of items on the Cognitive Complaint Index (CCI);
* depression severity: MADRS (Montgomery-Asberg Depression Rating Scale) ≥ 15;
* cognition: MOCA (Montreal Cognitive Assessment) ≥ 24;
* fluent in English;
* intact hearing / vision allowing completion of study procedures;
* for individuals on antidepressants at study entry, they must be on a stable dose for at least 6 weeks.

Exclusion Criteria:

* Other Axis I psychiatric disorders, except for anxiety symptoms occurring in a depressive episode;
* History of alcohol or drug dependence or abuse in the last 3 years;
* Tobacco or nicotine use in last year;
* History of a developmental disorder or IQ score < 70;
* Acute suicidality;
* Acute grief (<1 month);
* Current or past psychosis;
* Primary neurological disorder, including dementia, stroke, brain tumors, etc.;
* Any MRI contraindication;
* Unstable medical illness;
* Allergy or hypersensitivity to nicotine patches;
* Regular use of drugs with centrally acting cholinergic or anticholinergic properties in last 4 weeks, including acetylcholinesterase inhibitors;
* Current or planned psychotherapy;
* Electroconvulsive therapy (ECT) or transcranial magnetic stimulation (TMS) in last two months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Taylor, MD, MHSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gandelman JA, Kang H, Antal A, Albert K, Boyd BD, Conley AC, Newhouse P, Taylor WD. Transdermal Nicotine for the Treatment of Mood and Cognitive Symptoms in Nonsmokers With Late-Life Depression. J Clin Psychiatry. 2018 Aug 28;79(5):18m12137. doi: 10.4088/JCP.18m12137. PMID 30192444

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Nicotine Patch: Transdermal nicotine patch, administered on awakening and removed at bedtime (16h/d). Dosing began at 3.5mg patch/daily, titrated over study to maximum dose of 21mg patch/daily. Dose could be reduced to the prior level or an intermediate level for tolerability.
  Titration schedule: 3.5mg patch x 1 week, 7mg patch x 2 weeks, 14mg patch x 3 weeks, 21mg patch x 6 weeks.
  Nicotine: Open-label transdermal nicotine patch
Period: Overall Study
Arm/Group | Transdermal Nicotine Patch
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Past smoker (defined as smoking at least 1 cigarette daily for at least 6 months over the lifetime) [Count of Participants; unit: Participants] | 5
Depression severity (measured by Montgomery Asberg Depression Rating Scale total score) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician-rated measure of depression severity with a total score ranging from 0 to 60, where higher scores indicate greater depression severity.
  units on a scale | 27.7 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total MADRS (Montgomery Asberg Depression Rating Scale) Score
Description: Primary mood outcome measured by the total score of the clinician-rated MADRS. MADRS was measured every 3 weeks (baseline, week 3, week 6, week 9, and week 12). MADRS total score range is 0-60, where higher scores indicate greater depression severity.
Time Frame: Baseline to week 12
Population: Analyses included all participants, including the one subject who withdrew early. Missing values were imputed using the mean value of the sample at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 15
units on a scale | -18.45 (7.98)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p < 0.001, Regression, Linear; For change in depression severity (MADRS) over time, we used a linear mixed effects model with autoregressive of order 1 (AR(1)) temporal process

2. Primary Outcome: Change in Continuous Performance Task (CPT) Performance
Description: Primary cognitive outcome, the CPT is a neuropsychological test that measures attention. In this 14-minute test, participants are asked to respond when any letter appears, except the non-target letter "X". This test is conducted at baseline and at week 12. The specific primary outcome metric is standard error of change in the inter-stimulus hit reaction time, or variability between different trials. There is no absolute range, but lower scores indicate decreased variability across trials and overall better performance.
Time Frame: Baseline to week 12
Population: Subject who withdrew early not included due to no 12-week data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
milliseconds | -0.003 (0.135)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.761, Wilcoxon (Mann-Whitney); Wilcoxon signed-rank test

3. Secondary Outcome: Change in Snaith-Hamilton Pleasure Scale (SHAPS) Score
Description: Secondary mood outcome: Change in anhedonia measured by SHAPS, a self-report questionnaire that ranges from 0-42, where higher scores indicate greater anhedonia.
Time Frame: Baseline to week 12
Population: One subject not included due to early withdrawal
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
units on a scale | -3.4 (6.6)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Wilcoxon signed-rank test assessing for change from baseline to 12-weeks; Test type: Other; p = 0.084, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Penn State Worry Questionnaire (PSWQ)
Description: Secondary mood outcome: Change in anxiety and worry measured by PSWQ, a self-report questionnaire with a range of 16-80, where higher scores indicate greater anxiety and worry.
Time Frame: Baseline to week 12
Population: One participant not included due to early withdrawal.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
units on a scale | -5.1 (13.4)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Wilcoxon signed-rank test assessing for change from baseline to 12-weeks; Test type: Other; p = 0.073, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Ruminative Response Scale Total Score
Description: Secondary mood outcome: Change in rumination measured by the Ruminative Response Scale total score measured at baseline and week 12. This is a self-report scale with a range of 0-66, where higher scores indicate higher levels of rumination.
Time Frame: Baseline to week 12
Population: Subject who withdrew early not included due to no 12-week data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
units on a scale | -9.0 (10.0)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney); Wilcoxon signed-rank test

6. Secondary Outcome: Change in Apathy Evaluation Scale (AES)
Description: Secondary Mood Outcomes: Change in apathy as measured by the self-report AES, a questionnaire with a range of 0-54, where lower scores indicate greater apathy.
Time Frame: Baseline to 12 weeks
Population: Subject who withdrew early not included due to no 12-week data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
units on a scale | 7.7 (5.4)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

7. Secondary Outcome: Change in MFQ (Memory Frequency Questionnaire) Score
Description: Secondary cognitive outcome: Change in subjective cognitive performance as measured by MFQ, a self-report scale ranging from 64-448. Higher scores indicate better subjective memory function, while lower scores indicate poorer subjective memory function.
Time Frame: Baseline to week 12
Population: Subject who withdrew early not included due to no 12-week data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
units on a scale | 23.64 (40.96)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.049, Wilcoxon (Mann-Whitney); Wilcoxon signed-rank test

8. Secondary Outcome: Change in Choice Reaction Time (CRT) Performance
Description: Secondary cognitive outcome, a neuropsychological test measure of attention. We examined the total response time for the CRT. Lower scores indicate better performance.
Time Frame: Baseline to week 12
Population: Subject who withdrew early not included due to no 12-week data.
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
milliseconds | -16.0 (85.9)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.502, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

9. Secondary Outcome: Change in One-back Test Performance
Description: Secondary cognitive outcome examining change in speed of responses ton the one-back test, no absolute range. In this variant of the "N-back" task, participants view a series of cards, and indicate whether the card they are currently viewing is identical to the previously viewed card. Lower scores indicate better performance.
Time Frame: Baseline to week 12
Population: Subject who withdrew early not included due to no 12-week data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
milliseconds | -0.040 (0.065)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.049, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

10. Secondary Outcome: Change in NYU (New York University) Paragraph Recall Performance
Description: Secondary cognitive outcome of a neuropsychological test examining episodic memory performance using the NYU Paragraph Recall test. No absolute range. Higher scores indicate better performance.
Time Frame: Baseline to week 12
Population: Subject who withdrew early not included due to no 12-week data.
Measure: Mean (Standard Error); unit: Items correct
Arm/Group | Transdermal Nicotine Patch
Number analyzed (Participants) | 14
Items correct | 3.4 (5.8)
Statistical Analysis 1: Comparison: Transdermal Nicotine Patch; Test type: Other; p = 0.068, Wilcoxon (Mann-Whitney); Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events collected through query of subjects about any new or worsening problems or side effects, conducted at each contact.
Arm/Group | Transdermal Nicotine Patch
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transdermal Nicotine Patch (N=15)
Nausea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 4 — Symptoms included feelings of dizziness or lightheadedness
Anxiety (Psychiatric disorders) | 3 — Increases in subjective anxiety or tension
Headache (Nervous system disorders) | 4 — New onset of headaches or worsening pre-existing headache problem
Vivid Dreams (Nervous system disorders) | 3 — Increase frequency / intensity of "vivid" or lifelike dreams
Patch site reaction (Skin and subcutaneous tissue disorders) | 3 — Rash or pruritus at site where nicotine patch was applied

LIMITATIONS AND CAVEATS:
Open label trial design Only 8/14 participants who completed the study could tolerate the maximum patch dose of 21mg. The other 6 could only tolerate a maximum dose of 10.5mg, primarily due to adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT02816138/Prot_SAP_000.pdf